CLINICAL TRIAL: NCT02885168
Title: Modulation of Vasoreactivity in Septic Shock: Impact of Recombinant Protein C
Acronym: PCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-002319-16
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Septic Shock
Keywords: vasoreactivity; recombinant activated protein C
MeSH Terms: conditions — Shock, Septic | interventions — 3K3A-APC protein; drotrecogin alfa activated; Spectroscopy, Near-Infrared; Phenylephrine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shock + Treatment (Experimental): Patients treated with activated protein C
  Interventions: Drug: Recombinant Activated Protein C; Device: Near-infrared spectroscopy (NIRS); Drug: Phenylephrine; Biological: Blood sample
- Shock (Other): Patients not treated with activated protein C
  Interventions: Device: Near-infrared spectroscopy (NIRS); Drug: Phenylephrine; Biological: Blood sample

INTERVENTIONS:
Drug: Recombinant Activated Protein C — 24 μg/kg/h during 96 hours - intravenous injection
  Other Names: Xigris
  Arms: Shock + Treatment
Device: Near-infrared spectroscopy (NIRS) — After baseline measurement, cuff is blown up to obtain a muscular saturation at 40% and then deflated. Reactive hyperthermia is measured. It is considered as an index for endothelial function.
Drug: Phenylephrine — Continuous administration of phenylephrine with electric syringe with increasing dosing levels: 0.0; 0.02; 0.05; 0.1; 0.2; 0.5; 0.75; 1.00; 1.50; 3.00; 4.50; 6.00; 9.00 et 12 µg/kg/min. Each level is maintained for 5 minutes. Administration of phenylephrine is stopped progressively with the same schema.
  Arterial tension through an invasive approach is measured during the test.
Biological: Blood sample — Analysis of inflammation and cellular adhesion markers and free radicals

SUMMARY:
The purpose is to demonstrate that vasoreactivity of patients with septic shock evaluated with dose-response curve is diminished in septic shock and ameliorated by activated protein C (APC).

This amelioration is correlated to decrease of inflammation, decrease of reactive oxygen species (ROS) markers and increase of circulating catecholamines.

ELIGIBILITY:
Inclusion Criteria:

- Patients with septic shock as determined by standard criteria (including infection and severe infection)

Exclusion Criteria:

* Pregnant women
* Absence of signed informed consent. Due to gravity of medical situation of patients, inclusion will be possible after informed consent of a family member. As soon as possible, an informed consent will be obtained by patient
* Contraindication to Xigris: evolutive internal bleeding , intracranial pathology, neoplasia or brain involvement, concomitant heparin therapy >= 15 IU/kg/h, known hemorrhagic diathesis except acute coagulopathy subsequent to sepsis, severe chronic liver disease, platelet count < 30000 x 10^6/L, high bleeding risk, known hypersensibility to drotrecogin alfa (activated), one of excipients or bovine thrombin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Vascular reactivity measured with dose-response to phenylephrine | baseline
Vascular reactivity measured with dose-response to phenylephrine | 4 hours
Vascular reactivity measured with dose-response to phenylephrine | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LEVY, Principal Investigator — Réanimation Médicale - Hôpital de Brabois - CHRU Nancy

IPD SHARING:
Plan to Share IPD: No